CLINICAL TRIAL: NCT02105116
Title: AML Therapy With Irradiated Allogeneic Cells
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients were eligible to receive the experimental component of the protocol therapy.
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Roger Strair, MD, PhD, Professor of Medicine, RWJMS, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2013002693; NCI-2013-02408 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2013002693 (Other: IRB number); 021208 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — fludarabine phosphate; Cytarabine; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standard chemotherapy followed by allogenic therapy (Experimental): INDUCTION CHEMOTHERAPY: Patients receive standard induction chemotherapy with fludarabine phosphate IV over 1 hour QD for 5 days and cytarabine IV over 4 hours for 5 days. G-CSF 5 mcg/kg will be started at day14 if day14 bone marrow does not have >5% leukemic blasts. Treatment may continue for 1 or 2 courses at the discretion of the treating physician. If the patient enters a complete remission they are eligible for ALLOGENEIC CELLULAR THERAPY: Patients eligible for the experimental therapy undergo irradiated Donor Lymphocyte Infusion (DLI) of 3 x 10^8 CD3+ cells/kg at 8 weeks. Patients with stable disease may repeat irradiated DLI every 8-12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fludarabine phosphate; Drug: cytarabine; Biological: donor lymphocytes; Other: laboratory biomarker analysis; Drug: G-CSF

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Biological: donor lymphocytes — Undergo infusion of donor lymphocytes
Other: laboratory biomarker analysis — Correlative studies
Drug: G-CSF — Given IV
  Other Names: Filgrastim; Neupogen®

SUMMARY:
This pilot clinical trial studies if cells donated by a close genetic relative can help maintain acute myeloid leukemia (AML) complete remission (CR). Eligible patients will receive a standard induction chemotherapy. If a complete remission results they will receive irradiated allogeneic cells from a HLA haploidentical relative. Only patients who obtain a CR after the standard induction chemotherapy are eligible for the experimental therapy (irradiated haploidentical cells).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Toxicity of haploidentical allogeneic cellular therapy in patients in complete remission (CR) (or CR with incomplete platelet recovery [CRp]) after induction chemotherapy with fludarabine (fludarabine phosphate)-cytarabine.

II. Efficacy of haploidentical allogeneic cellular therapy in patients in CR (or CRp) after induction chemotherapy with fludarabine-cytarabine (remission rates at 6, 12, 18, 24 months).

SECONDARY OBJECTIVES:

I. Immunologic parameters before and after haploidentical therapy: host anti-leukemia T cells; host regulatory T cells.

OUTLINE:

INDUCTION CHEMOTHERAPY: Patients receive fludarabine phosphate intravenously (IV) over 1 hour once daily (QD) for 5 days and cytarabine IV over 4 hours for 5 days. Treatment may continue for 1 or 2 courses at the discretion of the treating physician.

ALLOGENEIC CELLULAR THERAPY: Patients undergo irradiated donor lymphocyte infusion (DLI) of 3 x 10^8 cluster of differentiation (CD)3+ cells/kg at 8 weeks. Patients with stable disease may repeat irradiated DLI every 8-12 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-M3 AML:

  * Refractory/relapsed AML OR
  * Initial diagnosis of AML in patient >= 60 years old
* Total bilirubin =< 1.5 times upper limit of normal (ULN) institutional limits (unless Gilbert's disease)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional ULN
* Cardiac left ventricular ejection fraction (LVEF) >= 35%
* Serum creatinine =< 1.5 mg/dl
* Any organ dysfunction thought to be secondary to disease will be considered separately and the patient will be included at the investigators discretion
* Patients must give informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* Must have a potential haploidentical donor (parent, sibling, child)
* A patient is eligible for second enrollment (allo-cellular therapy) if all of the following inclusion criteria are met:
* Patient must have documented CR or CRp after 1 or 2 cycles of fludarabine + cytarabine
* Patient must not be a candidate for an allo-hematopoietic stem cell transplant (HSCT)
* Patient must have a partially (>= 3/6 class I antigen) human leukocyte antigen (HLA)-matched (by serology or low resolution deoxyribonucleic acid [DNA] testing) relative able to serve as a donor
* Patients must not have active uncontrolled infections, other medical or psychological/social conditions that might increase the likelihood of patient adverse effects or poor outcomes
* Total bilirubin < 1.5 times upper limit of normal (ULN) institutional limits (unless Gilbert's disease)
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional ULN
* Serum creatinine < 2.0 mg/dl
* ECOG performance status =< 2
* DONOR: donor must be related to patient and be partially (>= 3/6 antigen) HLA-matched
* DONOR: donor must meet all New Brunswick Affiliated Hospitals (NBAH) requirements for hematopoietic stem cell donation, including:
* DONOR: age >= 18 years old
* DONOR: white blood cells (WBC) 4.0-10.0 x 10^3/mm^3
* DONOR: platelet count 150,000 to 440,000/mm^3
* DONOR: hemoglobin/hematocrit; 12.5-18 g/dl, 38 to 54%
* DONOR: not pregnant or lactating
* DONOR: not human immunodeficiency virus (HIV)-1, HIV-2, hepatitis C virus (HCV), hepatitis B core or human T-lymphotropic virus (HTLV)-I/II seropositive; hepatitis B surface antigen (HB S ag) (-); meet other infectious disease screening criteria utilized by NBAH Blood Center
* DONOR: no uncontrolled infections, other medical or psychological/social conditions, or medications that might increase the likelihood of patient or donor adverse effects or poor outcomes
* DONOR: meet other blood bank criteria for blood product donation (as determined by NBAH Blood Center screening history and laboratory studies)

Exclusion Criteria:

* History of current or prior medical problems that the investigator feels will prevent administration of therapy or assessment of response due to excess toxicity
* Patients with known active central nervous system (CNS) leukemia will be excluded from this clinical study
* Known HIV-positive patients are excluded from the study
* Patients may not be pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12-16 (Actual); Study Completion 2015-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the Rutgers Cancer Institute of New Jersey. The study was open to accrual on 02/17/2014 and was closed to accrual on 08/25/2015. The study was terminated on 12/16/2015.
Pre-assignment Details: We are reporting results on 6 eligible patients. One patient was deemed ineligible.
Groups:
- Treatment (Combination Chemotherapy, DLI): INDUCTION CHEMOTHERAPY: Patients receive fludarabine phosphate IV over 1 hour QD for 5 days and cytarabine IV over 4 hours for 5 days. G-CSF 5 mcg/kg will be started at day14 if day14 bone marrow does not have >5% leukemic blasts. Treatment may continue for 1 or 2 courses at the discretion of the treating physician.
  ALLOGENEIC CELLULAR THERAPY: Patients undergo irradiated Donor Lymphocyte Infusion (DLI) of 3 x 10^8 CD3+ cells/kg at 8 weeks. Patients with stable disease may repeat irradiated DLI every 8-12 weeks in the absence of disease progression or unacceptable toxicity.
  fludarabine phosphate: Given IV
  cytarabine: Given IV
  donor lymphocytes: Undergo infusion of donor lymphocytes
  laboratory biomarker analysis: Correlative studies
  G-CSF: Given IV
Period: Overall Study
Arm/Group | Treatment (Combination Chemotherapy, DLI)
Started | 6
Completed | 0
Not Completed | 6
Not completed — not eligible for step 2 of trial | 5
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Combination Chemotherapy, DLI)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Related to Experimental Therapy
Description: Patients will be observed for incidence of adverse events related to experimental therapy, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
  Of the 6 patients enrolled, all were ineligible to enter the experimental treatment phase of the study because of failure to reach complete remission. None of the enrolled patients received experimental therapy (allogeneic donor lymphocyte therapy). The one death occurred while receiving standard therapy prior to eligibility for experimental allogeneic therapy. The remained of patients were ineligible for experimental therapy because they did not obtain a complete remission after standard induction chemotherapy.
Time Frame: Up to 2 years
Arm/Group | Treatment (Combination Chemotherapy, DLI)
Number analyzed (Participants) | 0

2. Primary Outcome: Response Rate, Determined by Allogeneic Cell Therapy-related Mortality
Description: Patients' response rate will be determined by allogeneic cell therapy-related mortality. Of the 6 patients enrolled, all were ineligible to enter the experimental treatment phase of the study for failure to reach complete remission. Hence no outcomes are available.
Time Frame: Up to 2 years
Arm/Group | Treatment (Combination Chemotherapy, DLI)
Number analyzed (Participants) | 0

3. Primary Outcome: Response Rate, Determined by Duration of Complete Remission
Description: Patients will be scored as being in continuous remission at 2 years or having relapsed sooner. Of the 6 patients enrolled, all were ineligible to enter the treatment phase of the study for failure to reach complete remission for allogenic treatment.
Time Frame: Up to 2 years
Arm/Group | Treatment (Combination Chemotherapy, DLI)
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival Probability for CR
Description: Calculated using Kaplan-Meier estimation method. Corresponding 95% confidence interval will be provided. Of the 6 patients enrolled, all were ineligible to enter the experimental treatment phase of the study for failure to reach complete remission. Hence no outcomes are available.
Time Frame: At 2 years
Arm/Group | Treatment (Combination Chemotherapy, DLI)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 340 days per patient.
Arm/Group | Treatment (Combination Chemotherapy, DLI)
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes